CLINICAL TRIAL: NCT02275598
Title: A Pilot Phase II Study To Assess The Efficacy Of Brentuximab Vedotin Administered Sequentially With ABVD Chemotherapy In Patients With Untreated Hodgkin Lymphoma.
Brief Title: Brentuximab Vedotin Followed by ABVD in Patients With Previously Untreated Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Massimo Federico, MD, Full Professor, University of Modena and Reggio Emilia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV-ABVD
Record Dates: First submitted 2014-10-08; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BV-ABVD (Experimental): Treatment will consist of two three-weekly doses of Brentuximab vedotin, followed by standard treatment, ABVD (3 o 6 cycles q4w).
  Interventions: Drug: Brentuximab vedotin; Drug: ABVD

INTERVENTIONS:
Drug: Brentuximab vedotin — 1.8 mg/kg, IV (in the vein) on day 1 of each 28 day cycle. Number of Cycles: 2
  Other Names: Adcetris
Drug: ABVD — Doxorubicin 25 mg/m2 IV, Bleomycin 10,000 units/m2 IV, Vinblastine 6 mg/m2 IV, Dacarbazine 375 mg/m2 IV on days 1-15 of each 28 day cycle. Number of Cycles: 3 or 6 according to initial disease stage.

SUMMARY:
The purpose of this study is to assess the efficacy of two three-weekly 1.8 mg/kg Brentuximab vedotin administrations in untreated patients with Hodgkin Lymphoma (HL).

DETAILED DESCRIPTION:
This is a multicenter pilot phase II trial assessing 2 administrations of Brentuximab vedotin followed by PET scan and subsequent standard treatment with ABVD ± Radiotherapy. 12 patients defined by inclusion and exclusion criteria will be enrolled in one year. All subjects will be followed for disease evaluation every 3 months for one year after end of therapy until disease progression, death, initiation of alternative therapy, withdrawal of consent, or end of study. For all study procedures patient will be assigned a Unique Subject Identifier (SID) number that will be used to identify the subject during the screening process and throughout study participation. A master log will be maintained of all consented subjects and will document all screening failures (i.e. subjects who are consented but do not meet study eligibility criteria). Study records such as case report forms (CRFs) may be maintained electronically and require the same security and confidentiality as paper. Clinical information will not be released without written permission of the subject/legal representative, except as specified in the informed consent form

ELIGIBILITY:
Inclusion Criteria:

* Previously-untreated patients with classical Hodgkin Lymphoma according to the World Health Organisation (WHO) classification
* Histologically confirmed CD30+ HL
* Stage IA, IIA, IIIA
* Absence of bulky disease
* FDG-PET at baseline
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life expectancy > 6 months.
* Age 18-70 years.
* Patients must be available for periodic blood sampling, study-related assessments, and management of toxicity at the treating institution.
* Females of childbearing potential must have a negative pregnancy test result within three days of enrollment. All patients must agree to use effective contraceptive methods (one for male and two for female) during the course of the study and for 6 months following the end of full treatment (Brentuximab vedotin + ABVD +/- Radiotherapy).
* Written informed consent.
* Required baseline laboratory data:

Absolute neutrophil count ≥ 1000/μl Platelet count ≥ 50.000/ μl Serum bilirubin ≤ 1.5 times ULN Serum creatinine ≤ 1.5 times ULN Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN

Exclusion Criteria:

* Peripheral neuropathy > Grade 1
* Histologic diagnosis different from Hodgkin Lymphoma
* Compressive symptoms
* Patients previously treated with any anti-CD30 antibody
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive, or known or suspected infection active hepatitis C
* Patients with signs or symptoms of progressive multifocal leukoencephalopathy (PML)
* Patients with known cerebral/meningeal disease.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Complete Metabolic Response by FDG-PET | between day +8 and day +15 from second administration of Brentuximab
  Complete Metabolic Response will be defined by Deauville score 1, 2, 3.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 4 weeks from the end of full treatment program.
Progression Free Survival (PFS) | at 1 year from the end of full treatment program.
Number of Participants with Adverse Events | from C1D1 of Brentuximab vedotin up to 1 year from the end of full treatment program.
  All serious and on-serious adverse events will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, MD, Study Chair — Department of Diagnostic, Clinical and Public Health Medicine
Locations (3):
- Italy (3):
  - Institute of Hematology and Medical Oncology "L. e A. Seràgnoli" at the University of Bologna, Bologna
  - Department of Diagnostic, Clinical and Public Health Medicine, University of Modena and Reggio Emilia, Modena
  - Hematology, Azienda Ospedaliera Arcispedale S.Maria Nuova IRCCS, Reggio Emilia